CLINICAL TRIAL: NCT06029465
Title: Analyzing Engagement Trends in Rhabdomyosarcoma Clinical Trials: A Study of Participation Patterns Among Those Affected by the Disorder
Brief Title: Analyzing Engagement Trends in Rhabdomyosarcoma Clinical Trials
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 84447609
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Rhabdomyosarcoma
Keywords: Rhabdomyosarcoma
MeSH Terms: conditions — Rhabdomyosarcoma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study seeks to delve into the firsthand experiences of patients diagnosed with rhabdomyosarcoma who partake in a separate clinical trial featuring a specific medical intervention. The primary emphasis will be on meticulously tracking the rates of trial completion and withdrawal among these individuals.

The data collected from this study will help improve future outcomes for all rhabdomyosarcoma patients as well as those in under-represented demographic groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rhabdomyosarcoma
* Considered reliable, able to understand, and willing to perform all study procedures
* Signed Written Informed Consent

Exclusion Criteria:

* Currently enrolled in, have completed or have discontinued from a clinical trial involving an investigational drug
* Is pregnant, breastfeeding or expecting to conceive within the projected duration of the study
* Any serious and/or unstable pre-existing medical disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rhabdomyosarcoma who are actively considering enrolling in an observational clinical study for said condition, but have not yet completed enrollment and randomization phases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of rhabdomyosarcoma patients who decide to enroll in a clinical trial | 3 months
Rate of rhabdomyosarcoma patients who remain in clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sparber-Sauer M, Ferrari A, Kosztyla D, Ladenstein R, Cecchetto G, Kazanowska B, Scarzello G, Ljungman G, Milano GM, Niggli F, Alaggio R, Vokuhl C, Casanova M, Klingebiel T, Zin A, Koscielniak E, Bisogno G. Long-term results from the multicentric European randomized phase 3 trial CWS/RMS-96 for localized high-risk soft tissue sarcoma in children, adolescents, and young adults. Pediatr Blood Cancer. 2022 Sep;69(9):e29691. doi: 10.1002/pbc.29691. Epub 2022 Apr 19. PMID 35441463
- [Background] Saulnier-Sholler G, Duda DG, Bergendahl G, Ebb D, Snuderl M, Laetsch TW, Michlitsch J, Hanson D, Isakoff MS, Bielamowicz K, Kraveka JM, Ferguson W, Carmeliet P, De Deene A, Gijsen L, Jain RK. A Phase I Trial of TB-403 in Relapsed Medulloblastoma, Neuroblastoma, Ewing Sarcoma, and Alveolar Rhabdomyosarcoma. Clin Cancer Res. 2022 Sep 15;28(18):3950-3957. doi: 10.1158/1078-0432.CCR-22-1169. PMID 35833850
- [Background] Leiner J, Le Loarer F. The current landscape of rhabdomyosarcomas: an update. Virchows Arch. 2020 Jan;476(1):97-108. doi: 10.1007/s00428-019-02676-9. Epub 2019 Nov 6. PMID 31696361

DOCUMENTS (1):
  • Informed Consent Form (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT06029465/ICF_000.pdf